CLINICAL TRIAL: NCT07056166
Title: Prospective Observational Study: Ultrasound Predictors of Difficulty in Performing Epidural Anesthesia for Labor in Pregnant Patients.
Brief Title: Ultrasound Predictors of Difficulty in Performing Epidural Anesthesia for Labor in Pregnant Patients.
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Other Study IDs: AOP3720
Record Dates: First submitted 2025-06-20; First posted 2025-07-09 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Epidural Catheterization
Keywords: Epidural analgesia; Pregnancy; Spinal ultrasound; Difficult epidural; Obstetric anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant patients undergoing epidural placement for labor analgesia
  Interventions: Procedure: epidural catheter; Procedure: spine ultrasonography

INTERVENTIONS:
Procedure: epidural catheter — Epidural catheter placement for labor analgesia
Procedure: spine ultrasonography — An ultrasound scan will be performed on the spine to identify anatomical characteristics of potential interest

SUMMARY:
This is a prospective observational study conducted at the University Hospital of Padua. The goal is to identify ultrasound markers that can help predict whether placing an epidural catheter during labor will be difficult. Pregnant women who request epidural analgesia will undergo a quick ultrasound scan of their lower back before the procedure. The study will collect information such as age, weight, height, and spinal anatomy, as well as ultrasound measurements. This information will be compared with how easy or difficult it was to place the epidural. The study does not involve any experimental treatment and uses standard care procedures already in place. There are no additional risks or costs for participants.

DETAILED DESCRIPTION:
This is a single-center, prospective observational study aimed at evaluating whether specific ultrasound measurements of spinal structures in pregnant women can predict technical difficulty in placing an epidural catheter during labor analgesia. All procedures performed are part of standard care and are routinely offered in the labor and delivery unit. Patients who consent to participate will undergo a lumbar ultrasound prior to epidural catheter placement. Data will be collected regarding anatomical and clinical characteristics, ultrasound findings, and procedural details. The study will run for two years or until the estimated sample size of 563 patients is reached. The results are intended to identify non-invasive predictors of challenging epidural placement, potentially improving patient safety and resource allocation.

ELIGIBILITY:
-Inclusion Criteria: Pregnant women aged ≥18 years Candidates for epidural catheter placement for labor analgesia Provided written informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult pregnant women (≥18 years old) admitted to the Labor and Delivery Unit at the University Hospital of Padua who are candidates for epidural catheter placement for labor analgesia. All participants must provide written informed consent. No specific exclusion criteria apply.
Sampling Method: Non-Probability Sample
Enrollment: 563 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Difficulty of epidural catheter placement | Periprocedural
  Defined as the need for more than one puncture attempt (exiting the skin with the needle) or the involvement of a second operator to successfully place the epidural catheter.

SECONDARY OUTCOMES:
Number of puncture attempts | Periprocedural
  Number of attempts required to successfully insert the epidural catheter.
(Predictor of difficult Epidural) Distance from skin to spinous process at epidural placement level | Periprocedural
  The distance measured in cm between the skin surface and the spinous process at the intended epidural insertion site, assessed using ultrasound scanning.
(Predictor of difficult Epidural) Distance between spinous processes | Periprocedural
  Measured in centimeters by ultrasound to assess interspinous space width.
(Predictor of difficult Epidural) Distance from skin to transverse process | Periprocedural
  Measured in centimeters by ultrasound to assess distance between skin and transverse process.
(Predictor of difficult Epidural) Patient age | Baseline
  Measured in years
(Predictor of difficult Epidural) Pre-pregnancy weight | Baseline
  Measured in kg
(Predictor of difficult Epidural) Current weight | Baseline
  Measured in kg
(Predictor of difficult Epidural) Body Mass Index (BMI) | Baseline
  Measured in kg/cm2
(Predictor of difficult Epidural) Palpability of spinous processes | Periprocedural
  Measured as "Yes", "Not completely", "No"
(Predictor of difficult Epidural) Previous spinal surgery | Baseline
  "Yes" or "No" variable. Accounting for any type of vertebral surgery
(Predictor of difficult Epidural) Presence of scoliosis | Baseline
  "Yes" or "No" variable.
(Predictor of difficult Epidural) Operator Experience | Periprocedural
  Operator related. Defined as the number of epidural catheter previously positioned

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided